CLINICAL TRIAL: NCT04559789
Title: Digital Cognitive Multidomain Alzheimer's Risk Velocity Study (DC-MARVEL)
Brief Title: Reducing Dementia Risk With Digital Health Coaching
Acronym: DC-MARVEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neurotrack Technologies, Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R44AG063672-01 (NIH); R44AG063672 (NIH)
Record Dates: First submitted 2020-09-11; First posted 2020-09-23 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Alzheimer Disease; Dementia; Mild Cognitive Impairment; Cognitive Decline
Keywords: Dementia prevention; Risk reduction; Multi-domain lifestyle intervention; Behavior change
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Participants are randomly allocated to either the intervention or control group at the beginning of the study
Who Masked: Investigator, Outcomes Assessor
Masking Description: All study investigators that collect or analyze data are blinded to the group assignment for all participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Lifestyle Intervention (Experimental): Participants randomized to the intervention arm will receive access to a digital intervention consisting of the MindMate cognitive health app and Neurotrack's personalized health coaching platform.
  Interventions: Behavioral: MindMate + Health Coaching
- Health Education (Active Comparator): Participants randomized to the control arm will receive digital health education materials that mirror the content in the app.
  Interventions: Other: Health Education

INTERVENTIONS:
Behavioral: MindMate + Health Coaching — The MindMate app is a digital multi-domain lifestyle intervention designed to address modifiable risk factors for dementia. The app will be augmented with digital health coaching provided by Neurotrack.
  Arms: Digital Lifestyle Intervention
Other: Health Education — Health education materials delivered electronically
  Arms: Health Education

SUMMARY:
The Digital Cognitive Multi-domain Alzheimer's Risk Velocity (DC MARVEL) study is a 2-year randomized controlled trial on dementia prevention. The purpose of this study is to determine the effect of a digital cognitive health program on dementia risk, cognitive function, and general health outcomes in middle age to older adults compared to a control group that receives health education.

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) is expected to affect 131 million people worldwide by 2050, but as many as 40% of these cases may be prevented by targeting modifiable risk factors such as diet, physical activity, cognitive engagement, and smoking. Neurotrack Technologies, Inc. will test the efficacy of a digital multi-domain lifestyle intervention with health coaching for cognitive health designed to change behaviors associated with increased risk for AD. This digital intervention addresses the challenge of scaling effective multi-domain lifestyle interventions for cognitive health and has the potential to improve risk behaviors, thereby reducing and/or delaying cognitive decline in older adults at risk for AD.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75
* BMI 18.5 - 39.9 kg/m2
* Fluent in English (written and spoken)
* A minimum of 2 of the following risk factors for AD from ANU-ADRI: High school education or less; Overweight, or class I or class II obese (BMI 25-39.9 kg/m2); History of diabetes; History of hypertension; History of high cholesterol; History of smoking; History of traumatic brain injury
* Maximum of 1 of the following protective factors for AD from ANU-ADRI: High level of physical activity; High fish consumption; High level of cognitive engagement
* Ability to send and receive text messages
* Own a smartphone, have a reliable internet connection, and willing to use email
* Ability to participate in light to moderate physical activity
* Willingness to be randomized

Exclusion Criteria:

* Physician diagnosis of: mental health condition (e.g., eating disorder, alcohol/substance use, schizophrenia, etc.); neurologic conditions (e.g. epilepsy, stroke, multiple sclerosis, Parkinson's disease, brain tumor, or severe traumatic brain injury); dementia, probable dementia, or mild cognitive impairment; other significant health condition (e.g. congestive heart failure, chronic obstructive pulmonary disease, coronary artery disease, renal failure, chronic kidney disease, pulmonary hypertension)
* Recent cardiovascular event or recent treatment for cancer (within the last year); on dialysis; or on active organ transplant list
* Visual problems that prevent viewing screen at a normal distance (e.g., legal blindness, detached retina, occlusive cataracts)
* History of learning disability
* Currently participating in a formal cognitive training coaching program or other lifestyle change program (e.g. diabetes prevention program)
* Currently pregnant or planning on becoming pregnant in the next two years

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Composite dementia risk | Baseline to 24 months
  Change in dementia risk as determined by Australian National University Alzheimer's Disease Risk Index (ANU-ADRI). Scores range from -13 to 64, with higher scores representing a higher risk for dementia.

SECONDARY OUTCOMES:
Rate of cognitive decline | Baseline to 24 months
  Change in rate of cognitive decline as determined by Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). Scores range from 40-160, with higher scores representing better cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Glenn, PhD, Principal Investigator — Neurotrack Technologies, Inc.
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Myers JR, Bryk KN, Madero EN, McFarlane J, Campitelli A, Gills J, Jones M, Paulson S, Gray M, Glenn JM. Initial Perspectives From Rural-Residing Adults on a Digital Cognitive Health Coaching Intervention: Exploratory Qualitative Analysis. JMIR Form Res. 2024 Jul 22;8:e51400. doi: 10.2196/51400. PMID 39038282
- [Derived] Campitelli A, Paulson S, Gills JL, Jones MD, Madero EN, Myers J, Glenn JM, Gray M. A Novel Digital Digit-Symbol Substitution Test Measuring Processing Speed in Adults At Risk for Alzheimer Disease: Validation Study. JMIR Aging. 2023 Jan 27;6:e36663. doi: 10.2196/36663. PMID 36705951
- [Derived] Gray M, Madero EN, Gills JL, Paulson S, Jones MD, Campitelli A, Myers J, Bott NT, Glenn JM. Intervention for a Digital, Cognitive, Multi-Domain Alzheimer Risk Velocity Study: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Feb 4;11(2):e31841. doi: 10.2196/31841. PMID 35119374